CLINICAL TRIAL: NCT05027256
Title: Entia Liberty: Usability Validation
Status: Completed | Type: Observational
Sponsor: Entia Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 304701
Record Dates: First submitted 2021-08-26; First posted 2021-08-30 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Entia Liberty — Home Monitoring solution

SUMMARY:
This study forms part of Entia's clinical evidence for regulatory submission. This study evaluates Entia Liberty's validation of the device. Participants will be trained to take an Entia Liberty test in a simulated home environment and a trained healthcare professional will perform another test from the same participant (different finger) on a separate device. The results will be compared. Usability data will be observed and the participants will complete a questionnaire after the tests have been performed.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old at the time of study entry
* Can provide written informed consent
* Patients who are currently receiving standard of care systemic anti-cancer therapy (chemotherapy, immunotherapy, endocrine and targeted therapy) for solid organ malignancy and have received at least one cycle
* Sufficient hearing to be able to participate in a video training session

Exclusion Criteria:

* Known inherited or acquired bleeding disorder
* History of haematological malignancy
* Known poorly controlled anti-coagulation
* Inadequate use and understanding of the English language, requiring a translator
* Participant unlikely to be able to perform fine manipulation required to use lancet or cartridge to obtain capillary blood sample and result
* Previously taken part in the 'PERTH-2' study involving a prototype device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants recruited from the outpatients clinic at the Christie
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Number of participants able to use the Entia Liberty device as specified in the validation procedure is 80%. | 3 months
  At least 24 of the participants are able to complete the Entia Liberty test.
Number of participants with new severe usability problems identified. | 3 months
  Identification of the number of participants that were deviating away from the instructions for use, resulting in increased risk to the results or themselves
Number of participants with study-related adverse events as assessed by the Residual Risk analysis of the usability data using predefined criteria for severity and occurrence in accordance with ISO 14971:2019(E) | 3 months
  Residual Risk analysis of the usability data using predefined criteria for severity and occurrence in accordance with ISO 14971:2019(E)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Buckinghamshire Healthcare NHS Trust, Aylesbury
  - The Christie NHS Foundation Trust, Manchester